CLINICAL TRIAL: NCT01965639
Title: A Clinical Intervention to Serve High-Risk Patients in the Southeastern Diabetes Initiative and Durham Diabetes Coalition
Brief Title: Southeastern Diabetes Initiative Clinical Intervention
Acronym: SEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00043463; 1C1CMS331018 (Other Grant/Funding Number: Centers for Medicare and Medicaid Services)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; Standard of care; Quality of life; Disease management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Risk group (Experimental): Extension of Care
  Interventions: Other: Extension of Care

INTERVENTIONS:
Other: Extension of Care — Clinical care will be delivered by a multidisciplinary team including (but not limited to) a physician, nurse practitioner, dietitian, pharmacist, licensed clinical social worker (LCSW), case manager, health educator and a community health worker in community settings including home visits and community based clinics.

SUMMARY:
The purpose of the Southeastern Diabetes Initiative Clinical Intervention is to augment existing standard of care in an effort to (1) improve population level diabetes management, health outcomes and quality of life for diagnosed and undiagnosed adults living with Type 2 Diabetes Mellitus, (2) reduce disparities in diabetes management, health outcomes and quality of life for adults living with Type 2 Diabetes Mellitus, and (3) reduce healthcare costs associated with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Clinical care will be delivered by a multidisciplinary team including (but not limited to) an physician, nurse practitioner, dietician, pharmacist, licensed clinical social worker (LCSW), case manager, health educator and a community health worker. Care will be delivered in community settings including home visits and community based clinics. With the exception of specific surveys (listed in the Study Intervention section) all data are being collected for the purpose of delivery of standard preventive care and clinical care. The population group will include patients diagnosed with Type 2 Diabetes Mellitus in four Southern United States counties, meeting certain inclusion criteria, and deemed "high risk" as determined by a set of standard criteria or a risk algorithm run on secondary data.

The investigators plan to characterize patients diagnosed or at risk for diabetes mellitus, and allow more detailed knowledge of their health than is provided by standard public health data. The investigators will use descriptive, parametric and non-parametric statistics to describe baseline characteristics (demographics and clinical measures of disease severity) of the sample and will compare responders and dropouts on independent and dependent variables, report any significant differences, and include this in the interpretation of results.

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18yrs
* Diagnosis of Type 2 diabetes
* Reside in Durham County, NC, Cabarrus County, NC, Quitman County, MS or Mingo County, WV or the neighboring areas and receive the majority of their healthcare in the four listed counties.
* Have capacity to give consent (or have a surrogate legally authorized representative or caregiver provide consent on their behalf).
* Defined as high risk by the risk algorithm or their primary care clinician.
* Referral from the primary care clinician or patient's medical home if one has been designated.

Exclusion Criteria:

* Lack capacity to make decisions and do not have a surrogate with authority to make health care decisions.
* Have a terminal illness with a life expectancy of 6 months or less
* Diagnosis of Type 1 diabetes or gestational diabetes
* Currently pregnant (confirmed via self-report and/or medical record)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2013-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 24 months

SECONDARY OUTCOMES:
Rate of health services utilization | up to 24 months
  As measured by inpatient hospital admissions and emergency department visits
Change in Medication Adherence | Baseline, 6, 12, 18, and 24 months
  As measured by the Morisky Medication Adherence Score
Change in HbA1c | Baseline, 6, 12, 18, and 24 months
Change in blood lipids | Baseline, 6, 12, 18, and 24 months
  Measurements include total cholesterol, HDL, LDL, triglycerides
Change in blood glucose | Baseline, 6, 12, 18, and 24 months
Change in blood pressure | Baseline, 6, 12, 18, and 24 months
Incidence of micro- and macro-vascular complications | Up to 24 months
  Includes retinopathy, neuropathy, kidney disease, cardiovascular disease
Change in patient-reported outcomes | Baseline, 6, 12, 18, and 24 months
  Includes results from PHQ 2, PAM-13, PROMIS 9, and REALM-SF surveys

CONTACTS AND LOCATIONS:
Overall Officials: Robert Califf, MD, Principal Investigator — Duke Translational Medicine Institute; Bryan Batch, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Mississippi Public Health Institute, Madison, Mississippi
  - Durham County Department of Public Health, Durham, North Carolina
  - Cabarrus Health Alliance, Kannapolis, North Carolina
  - Williamson Health and Wellness Center, Williamson, West Virginia